CLINICAL TRIAL: NCT05762835
Title: Virtual Family-Centered Rounds in the Neonatal Intensive Care Unit: a Cluster Randomized Controlled Trial
Brief Title: Neonatal Intensive Care Unit Virtual Family-Centered Rounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1764454
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Disorder; Neonatal Disease
Keywords: Pediatrics; Neonatal Intensive Care Units; Neonate; Clinical Trial; Telemedicine; Patient-Centered Care; Patient Reported Outcome Measures
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Virtual Family-Centered Rounds [FCR]) (Experimental): Virtual FCR-arm parents/guardians (referred to as "parents" hereafter) will have the option use have the option to use telehealth for virtual rounds. Parents can participate in virtual FCR as much, or as little, as they choose. Parents also will have the option to attend FCR in person or to not attend FCR.
  Interventions: Behavioral: Virtual family-centered rounds (FCR)
- Control (Usual Care) (No Intervention): Usual care-arm parents will receive usual care. Usual care-arm parents will have the option to attend FCR in person or to not attend FCR.

INTERVENTIONS:
Behavioral: Virtual family-centered rounds (FCR) — Parents will be given the option to join FCR virtually or in-person; this intervention is changing the behavior of how providers deliver healthcare and how parents engage in their child's care.
  The NICU team members will use a computer with a speaker and pan-tilt-zoom camera, mounted on a stand with wheels to launch telehealth connections using the secure application called ExtendedCare. From within this telehealth connection, a NICU team member will send an electronic message (e.g. via text or email) to the subscribed parent(s) and wait for the parent to join the visit to establish a secure videoconference. The message to the parent includes a link that can be clicked to open a browser that allows the parent to join the telehealth visit. FCR will then proceed in usual fashion with the NICU team members and - if in attendance - parent(s).
  Arms: Intervention (Virtual Family-Centered Rounds [FCR])

SUMMARY:
The aim of this study is to evaluate the impact of virtual family-centered rounds in the neonatal intensive care unit on parental and neonatal outcomes.

ELIGIBILITY:
Enrolling family units (which consists of INFANTS and PARENTS [SURVEYS]):

INFANT Inclusion

* Infants aged less than 365 days who are admitted to the NICU
* Have at least one adult parent or guardian with English proficiency

INFANT Exclusion

* Have restrictions placed by child protective services, including visitation restrictions or restricted access to patient information
* Infants with a previous NICU admission (and enrollment) during the trial period

PARENTS [SURVEYS] Inclusion

* Parents/guardians of the eligible infants (described above)
* Age 18 years and older

PARENTS [SURVEYS] Exclusion

* Age less than 18 years
* Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Rosenthal, MD, MAS, Principal Investigator — University of California, Davis
Locations (1):
- The Regents of the University of California, Davis, Sacramento, California, United States

REFERENCES:
- [Derived] Rosenthal JL, Tancredi DJ, Marcin JP, Ketchersid A, Horath ET, Zerda EN, Bushong TR, Merriott DS, Romano PS, Young HM, Hoffman KR. Virtual family-centered hospital rounds in the neonatal intensive care unit: protocol for a cluster randomized controlled trial. Trials. 2023 May 16;24(1):331. doi: 10.1186/s13063-023-07340-x. PMID 37194089
- [Derived] Rosenthal JL, Tancredi DJ, Marcin JP, Ketchersid A, Horath ET, Zerda EN, Bushong TR, Merriott DS, Romano PS, Young HM, Hoffman KR. Virtual Family-Centered Rounds in the Neonatal Intensive Care Unit: Protocol for a Cluster Randomized Controlled Trial. Res Sq [Preprint]. 2023 Apr 17:rs.3.rs-2644794. doi: 10.21203/rs.3.rs-2644794/v1. PMID 37131689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Family units enrolled and randomized. At time of enrollment, the number of infants was known, but the number of parents was unknown (because at that time did not know if family units had 1 vs. 2 parents/guardians). Enrolled 486 families (514 infants).
Units Other Than Participants: families
Groups:
- Intervention (Virtual Family-Centered Rounds [FCR]): Virtual FCR-arm parents/guardians (referred to as "parents" hereafter) will have the option use have the option to use telehealth for virtual rounds. Parents can participate in virtual FCR as much, or as little, as they choose. Parents also will have the option to attend FCR in person or to not attend FCR.
  Virtual family-centered rounds (FCR): Parents will be given the option to join FCR virtually or in-person; this intervention is changing the behavior of how providers deliver healthcare and how parents engage in their child's care.
  The NICU team members will use a computer with a speaker and pan-tilt-zoom camera, mounted on a stand with wheels to launch telehealth connections using the secure application called ExtendedCare. From within this telehealth connection, a NICU team member will send an electronic message (e.g. via text or email) to the subscribed parent(s) and wait for the parent to join the visit to establish a secure videoconference. The message to the parent includes a link that can be clicked to open a browser that allows the parent to join the telehealth visit. FCR will then proceed in usual fashion with the NICU team members and - if in attendance - parent(s).
Period: Overall Study
Arm/Group | Intervention (Virtual Family-Centered Rounds [FCR]) | Control (Usual Care)
Started | 345; 325 families (Family units enrolled and randomized. At time of randomization, the number of infants was known, but the number of parents was unknown (because at that time did not know if family units had 1 vs. 2 parents/guardians). Randomized 325 families (345 infants) to the intervention arm.) | 169; 161 families (Family units enrolled and randomized. At time of randomization, the number of infants was known, but the number of parents was unknown (because at that time did not know if family units had 1 vs. 2 parents/guardians). Randomized 161 families (169 infants) to the control arm.)
Completed | 342; 322 families (Outcomes data analyzed for 322 families (342 infants, 430 parents) in the intervention arm.) | 168; 160 families (Outcomes data analyzed for 160 families (168 infants, 219 parents) in the control arm.)
Not Completed | 3; 3 families | 1; 1 families

BASELINE CHARACTERISTICS:
Population: Overall # baseline participants is 322 intervention families (342 infants, 242 P1s, 188 P2s = 772 total) & 160 control families (168 infants, 119 P1s, 100 P2s = 387 total). Each family consisted of different #s of infants (e.g., twins) and different #s of parents (i.e., 1 to 2 parents/guardians per family) participants.
  Baseline data includes (a) enrolled infants plus (b) parents.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (Virtual Family-Centered Rounds [FCR]) | Control (Usual Care) | Total
Number analyzed (Participants) | 772 | 387 | 1159
Age, Categorical [Count of Participants; unit: Participants] — Population: Each family consisted of different #s of infants (e.g., twins/other multiples) and different #s of parents (i.e., 1 to 2 parents/guardians per family) participants. At time of randomization, the number of infants was known, but the number of parents was unknown (because at that time did not know if family units had 1 vs. 2 parents/guardians).
  Participants
    Participants: <=18 years | 342 | 168 | 510
    Participants: Between 18 and 65 years | 430 | 219 | 649
    Participants: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall number of baseline participants includes all individuals enrolled in the study (infants and their parents). Each baseline row reports data from a specific sub-population: infants, Parent 1s, and Parent 2s. The number analyzed in each row reflects the actual number of participants in that subgroup only.
  years
    Infants: number analyzed (Participants) | 342 | 168 | 510
    Infants | 0.01 (0.05) | 0.01 (0.04) | 0.01 (0.04)
    Parent 1: number analyzed (Participants) | 242 | 119 | 361
    Parent 1 | 31.1 (6.0) | 31.7 (5.6) | 31.3 (5.8)
    Parent 2: number analyzed (Participants) | 188 | 100 | 288
    Parent 2 | 33.5 (7.3) | 34.3 (7.3) | 33.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Parent participants included those with unknown sex
  Participants
    Infant: number analyzed (Participants) | 342 | 168 | 510
    Infant: Female | 154 | 68 | 222
    Infant: Male | 188 | 100 | 288
    Parent 1: number analyzed (Participants) | 242 | 119 | 361
    Parent 1: Female | 240 | 118 | 358
    Parent 1: Male | 2 | 1 | 3
    Parent 2: number analyzed (Participants) | 188 | 100 | 288
    Parent 2: Female | 11 | 3 | 14
    Parent 2: Male | 177 | 97 | 274
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 510 (infants) + 361 (parent 1) + 288 (parent 2) = 1159 total
  Participants
    Infant: number analyzed (Participants) | 342 | 168 | 510
    Infant: American Indian or Alaska Native | 3 | 1 | 4
    Infant: Asian | 27 | 18 | 45
    Infant: Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
    Infant: Black or African American | 36 | 10 | 46
    Infant: White | 138 | 61 | 199
    Infant: More than one race | 0 | 0 | 0
    Infant: Unknown or Not Reported | 138 | 76 | 214
    Parent 1: number analyzed (Participants) | 242 | 119 | 361
    Parent 1: American Indian or Alaska Native | 10 | 3 | 13
    Parent 1: Asian | 29 | 15 | 44
    Parent 1: Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
    Parent 1: Black or African American | 27 | 7 | 34
    Parent 1: White | 103 | 62 | 165
    Parent 1: More than one race | 22 | 9 | 31
    Parent 1: Unknown or Not Reported | 46 | 20 | 66
    Parent 2: number analyzed (Participants) | 188 | 100 | 288
    Parent 2: American Indian or Alaska Native | 4 | 4 | 8
    Parent 2: Asian | 24 | 12 | 36
    Parent 2: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    Parent 2: Black or African American | 14 | 7 | 21
    Parent 2: White | 89 | 56 | 145
    Parent 2: More than one race | 19 | 5 | 24
    Parent 2: Unknown or Not Reported | 36 | 16 | 52
Region of Enrollment [Number; unit: participants]
  United States | 772 | 387 | 1159

OUTCOME MEASURES:

1. Primary Outcome: Parent FCR Attendance
Description: Obtained from FCR weekday observations. Defined at family unit level, accounting for possibility of multiple enrolled infants per family and variable eligible FCR encounters for each infant. We will compute the total number of possible weekday FCR encounters per family ('denominator') and the number of those for which at least 1 parent is present virtually or in-person ('numerator'). The outcome measure will be reported as a proportion (numerator/denominator). For example, if a family has 2 infants, 1 whose NICU hospitalization included 5 eligible FCR encounters and another whose NICU hospitalization includes 7 eligible FCR encounters, that family will be counted as having twelve eligible FCR encounters ('denominator'). If at least 1 parent is present for 4 of the first infant's encounters and 6 of the second infant's encounters, the family would be counted as having attended 10 ('numerator') of the 12 eligible FCR encounters. The proportion for that family unit is 0.83.
Time Frame: Length of neonatal intensive care unit [NICU] stay (assessed up to 396 days)
Measure: Mean (95% Confidence Interval); unit: proportion of encounters
Arm/Group | Intervention (Virtual Family-Centered Rounds [FCR]) | Control (Usual Care)
Number analyzed (Participants) | 322 | 160
proportion of encounters | 0.56 [0.51 to 0.61] | 0.12 [0.09 to 0.16]

2. Secondary Outcome: Parent Experience
Description: Unit of measure: mean score; Measure/Tool: Emergency Department CAHPS (Consumer Assessment of Healthcare Providers and Systems) (parent survey, 2 items measuring overall experience).
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

3. Secondary Outcome: Family-Centered Care
Description: Unit of measure: mean score; Measure/Tool: Family-Centered Care Experience (FACCE) (parent survey)
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

4. Secondary Outcome: Parent Activation
Description: Unit of measure: mean score; Measure/Tool: Parent-Patient Activation Measure (P-PAM) (parent survey)
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

5. Secondary Outcome: Parent Health-related Quality of Life
Description: Unit of measure: mean score. Measure/Tool: PedsQL Family Impact Module (parent survey)
Time Frame: Day 0/30/60/90 (post-NICU discharge)
Reporting Status: Not Posted

6. Secondary Outcome: NICU Length of Stay
Description: Unit of measure: days in NICU. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

7. Secondary Outcome: Breastmilk Feeding
Description: Dichotomous outcomes. Include (a) breastmilk feeding initiation, (b) any breastmilk feeding at the time of discharge from the NICU (and 90 days later), and (c) exclusive breastmilk feeding at the time of discharge from the NICU (and 90 days later). Breastmilk feeding includes consuming milk from the birth parent via any delivery method (e.g., bottle, feeding tube, breast). Any breastmilk feeding will be defined as the infant consuming any amount of milk from the birth parent, with or without the addition of formula or fortifier. Exclusive breastmilk feeding will be defined as 100% of base feeding type as milk from the birth parent, with or without a bovine or human fortifier. Obtained from electronic health record (0 days) and parent survey (90 days).
Time Frame: Day 0/90 (post-NICU discharge)
Reporting Status: Not Posted

8. Secondary Outcome: Postnatal Growth Failure (Dichotomous)
Description: Measure/Tool: Sex-specific Fenton growth charts. This dichotomous outcome will define growth failure as a weight-for-gestational-age Z-score decline of more than 0.8 standard deviations (SD) from birth to discharge. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

9. Secondary Outcome: Postnatal Growth Failure (Categorical)
Description: Measure/Tool: Sex-specific Fenton growth charts. This categorical outcome will classify the degree of growth failure as none (no decline or a decline </=0.8 SD), mild (>0.8 and </=1.2 SD), moderate (>1.2 and </=2 SD), or severe (>2 SD). Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Neonatal Growth Velocity
Description: Continuous variable. Measure/Tool: Sex-specific Fenton growth charts. Calculate change in Z-score divided by number of days in the NICU. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Adverse Events and Errors
Description: Include the rates of harmful errors, non-harmful errors, and overall errors (harmful errors plus non-harmful errors). Obtained via review of data from electronic health record, incident report system, and solicited reports. Two neonatologists, blinded to the study arm, will independently categorize each event as a harmful error (preventable adverse event), non-harmful error, non-preventable adverse event, or exclusion.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: 30-day Revisit
Description: Defined as post-discharge revisits to any emergency department. Obtained from electronic health record and parent-reported survey.
Time Frame: Day 30 (post-NICU discharge)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: 30-day Readmission
Description: Defined as post-discharge unplanned readmissions to any hospital. Obtained from electronic health record and parent-reported survey.
Time Frame: Day 30 (post-NICU discharge)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Temperature Instability
Description: Dichotomous variable defined as any occurrence of a temperature below 36 degrees C during the NICU hospitalization. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Central Line-associated Bloodstream Infection
Description: Dichotomous variable defined as any occurrence during the NICU hospitalization of a laboratory-confirmed bacterial or viral bloodstream infection that develops with a central line in place and is not related to an infection at another site. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Central Line Days
Description: Number of days among the total number of NICU days that the infant has an umbilical catheter or one or more central lines in place. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Antibiotic Days
Description: Number of days among the total number of NICU days that the infant receives intramuscular or intravascular antibacterial or antifungal agents. Obtained from electronic health record.
Time Frame: Day 0 (post-NICU discharge)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 13 months
Description: Adverse event data were collected and monitored for infant participants only. Adverse events were not assessed or recorded for parent participants as part of the study's safety monitoring.
Arm/Group | Intervention (Virtual Family-Centered Rounds [FCR]) | Control (Usual Care)
All-Cause Mortality (participants affected / at risk) | 13/342 | 6/168
Serious Adverse Events (participants affected / at risk) | 0/342 | 0/168
Other Adverse Events (participants affected / at risk) | 0/342 | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT05762835/Prot_SAP_000.pdf